CLINICAL TRIAL: NCT04309877
Title: Pilot Randomized Controlled Trial of Theophylline for Attenuation of Lipopolysaccharide-Induced Depressive Symptoms
Brief Title: Theophylline for Depression Study
Acronym: T-DEP
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Hyong Jin Cho, Associate professor, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 20-000005
Record Dates: First submitted 2020-03-10; First posted 2020-03-16 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Lipopolysaccharides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PO theophylline & IV LPS (Experimental): Oral (PO) theophylline 400 mg/day for 2 weeks followed by a single intravenous (IV) bolus of lipopolysaccharide (LPS) 0.8 ng/kg of body weight
  Interventions: Drug: Theophylline ER; Biological: Lipopolysaccharide (LPS)
- PO placebo & IV LPS (Experimental): PO methylcellulose (placebo) daily for 2 weeks followed by a single intravenous (IV) bolus of lipopolysaccharide (LPS) 0.8 ng/kg of body weight
  Interventions: Other: PO placebo; Biological: Lipopolysaccharide (LPS)
- PO theophylline & IV placebo (Experimental): PO theophylline 400 mg/day for 2 weeks followed by a single IV bolus of 0.9% saline
  Interventions: Drug: Theophylline ER; Other: IV placebo
- PO placebo & IV placebo (Placebo Comparator): PO methylcellulose (placebo) daily for 2 weeks followed by a single IV bolus of 0.9% saline
  Interventions: Other: PO placebo; Other: IV placebo

INTERVENTIONS:
Drug: Theophylline ER — Capsules of theophylline ER
  Arms: PO theophylline & IV LPS; PO theophylline & IV placebo
Other: PO placebo — Capsules of methylcellulose
  Arms: PO placebo & IV LPS; PO placebo & IV placebo
Biological: Lipopolysaccharide (LPS) — Purified bacterial wall component as an inflammatory challenge
  Arms: PO placebo & IV LPS; PO theophylline & IV LPS
Other: IV placebo — Normal (0.9%) saline
  Arms: PO placebo & IV placebo; PO theophylline & IV placebo

SUMMARY:
Depression is very common and poses a huge disease burden. About 20% of the US population suffers from depression at least once in their lifetime. Inflammations that are hidden inside our body as a result of aging, obesity, chronic diseases, or certain treatments (e.g., interferon for hepatitis C) appear to cause depressive symptoms and even clinical depression. Individuals with such inflammations are more likely to suffer from depression and are less likely to respond to currently available antidepressant medications. This study will test theophylline, a medication currently used for asthma treatment, as a new way to mitigate depressive symptoms in response to such inflammations. This study begins with a 90-minute screening session to determine whether participants are eligible to join the main study. Those who meet the eligibility criteria will then join the main study, which will consist of taking theophylline or methylcellulose (i.e., oral placebo) for 2 weeks at home and an 8-hour session at the UCLA Medical Center. Approximately 20 healthy adults will be recruited for participation in the study. During the course of the study, participants will take theophylline or methylcellulose for 2 weeks at home and then will be injected either lipopolysaccharide (LPS) or saline (i.e., intravenous placebo) at the UCLA Medical Center. LPS is a bacterial substance that can initiate chemical reactions that are similar to those seen in individuals with mild sickness symptoms, such as a slight increase in body temperature, muscle aches, or tiredness. It is a safe way of investigating the body's response to inflammation and how these changes may alter cognitive, emotional, or neural function. It has been given thousands of times to healthy volunteers - both younger and older adults - without any serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* in good general health (as evaluated during the phone and in-person screening sessions)
* aged 18-65 years
* if female, using adequate birth control

Exclusion Criteria:

* history of hypersensitivity to xanthine derivatives (a contraindication to theophylline treatment)
* pregnant or planning to become pregnant in the next 6 months
* current breastfeeding
* chronic diseases such as cardiovascular disease, hepatic impairment, peptic ulcer disease, and seizure disorders
* current use of prescription medications such as steroids, non-steroid anti-inflammatory drugs, immune modifying drugs, opioid analgesics, and psychotropics
* Axis I psychiatric disorders including current major depressive disorder
* current depressive symptoms assessed by the Patient Health Questionnaire (PHQ-9 ≥ 5)
* heavy smoking (1 pack or more per day)
* excessive caffeine use (>600 mg/day)
* Body-mass index > 35 due to the effects of obesity on cytokine activity
* evidence of recreational drug use from urine test
* evidence of pregnancy from urine test
* evidence of clinically significant rhythm abnormality on a resting electrocardiogram (ECG)
* clinically significant abnormalities on screening laboratory tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in depressed mood from baseline | At baseline and then at 1, 1.5, 2, 3, 4, 5, and 6 hours after LPS (or saline) administration
  Short Form of the Profile of Mood States (POMS-SF) Depression Subscale with higher scores indicating more severe depressed mood (range 0-32)

SECONDARY OUTCOMES:
Change in tension/anxiety from baseline | At baseline and then at 1, 1.5, 2, 3, 4, 5, and 6 hours after LPS (or saline) administration
  Short Form of the Profile of Mood States (POMS-SF) Tension Subscale with higher scores indicating more severe tension/anxiety (range 0-24)
Change in depressive symptoms from baseline | At baseline and then at 2, 4, and 6 hours after LPS (or saline) administration
  Montgomery-Asberg Depression Rating Scale (MADRS): a clinician-rated questionnaire of depressive symptoms with scores ranging from 0 to 60, with higher scores indicating more severe depressive symptoms
Change in feelings of social disconnection from baseline | At baseline and then at 2, 4, and 6 hours after LPS (or saline) administration
  Feelings of Social Disconnection Scale: a self-report questionnaire of feelings of social disconnection with scores ranging from 0 to 28, with higher scores indicating more severe feelings of social disconnection
Change in fatigue from baseline | At baseline and then at 1, 1.5, 2, 3, 4, 5, and 6 hours after LPS (or saline) administration
  Short Form of the Profile of Mood States (POMS-SF) Fatigue Subscale with higher scores indicating more severe fatigue (range 0-20)
Change in confusion from baseline | At baseline and then at 1, 1.5, 2, 3, 4, 5, and 6 hours after LPS (or saline) administration
  Short Form of the Profile of Mood States (POMS) Confusion Subscale with higher scores indicating more severe confusion (range 0-20)
Change in verbal memory from baseline | At baseline and then 3 hours after LPS (or saline) administration
  Verbal memory measured using computerized tests from CNS Vital Signs™
Change in visual memory from baseline | At baseline and then 3 hours after LPS (or saline) administration
  Visual memory measured using computerized tests from CNS Vital Signs™
Change in executive function from baseline | At baseline and then 3 hours after LPS (or saline) administration
  Executive function measured using computerized tests from CNS Vital Signs™
Change in attention from baseline | At baseline and then 3 hours after LPS (or saline) administration
  Attention measured using computerized tests from CNS Vital Signs™

OTHER OUTCOMES:
Subjective Sensitivity to Social Rejection | 2 hours after LPS (or saline) administration
  Cyberball Social Exclusion Task
Negative Bias in Facial Emotion Recognition | 2 hours after LPS (or saline) administration
  Emotional Face Recognition Task
Reward | 2 hours after LPS (or saline) administration
  Reward Learning Task
Change in proinflammatory cytokines from baseline | At baseline and then at 1, 1.5, 2, 3, 4, 5, and 6 hours after LPS (or saline) administration
  Plasma proinflammatory cytokines (interleukin-1 receptor antagonist, interleukin-6, tumor necrosis factor-α, and soluble tumor necrosis factor receptor)
Change in kynurenine Metabolites from baseline | At baseline and then at 1, 1.5, 2, 3, 4, 5, and 6 hours after LPS (or saline) administration
  Plasma tryptophan, kynurenine, quinolinic acid, and kynurenic acid
Change in gene expression from baseline | At baseline and 30 minutes after LPS (or saline) administration
  Genome-wide transcriptional profiling with focus on the percentage increase from baseline to 30 minutes after LPS (or saline) administration in activities of transcription factors related to immune activation, sympathetic activation, and glucocorticoid insensitivity: respectively, nuclear factor kappa-B (NF-kB), cAMP response element-binding protein (CREB), and glucocorticoid receptor (GR).

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Cousins Center for Psychoneuroimmunology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No